CLINICAL TRIAL: NCT02408198
Title: The Street Smart Group: A Feasibility Trial of a Group Intervention Targeting Anxiety Processes in Paranoia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Amy Hardy, Research Clinical Psychologist, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R&D 2013/066
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Paranoia; Schizophrenia-spectrum Diagnosis
MeSH Terms: conditions — Paranoid Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate therapy (Experimental): Therapy will be delivered for a period of 6 weeks immediately after randomisation
  Interventions: Behavioral: Anxiety intervention
- Delayed therapy (No Intervention): Therapy will be delayed until 10 weeks following randomisation, and then delivered over a 6 week period

INTERVENTIONS:
Behavioral: Anxiety intervention — The intervention is based on a brief CBT for psychosis (CBTp) programme, focusing on understanding and managing anxiety processes that contribute to persecutory threat beliefs when in busy urban environments. The novel aspect of this intervention is that it is delivered in a group format. The intervention consists of six sessions which will be delivered on a weekly basis. Throughout the intervention there is an emphasis on setting tasks to practice applying the new skills outside of sessions, to help the person build confidence in being able to manage paranoia and feel less distressed in their daily life.
  Arms: Immediate therapy

SUMMARY:
This study aims to evaluate a novel group psychological intervention targeting anxiety triggered by urban environments for people with paranoia.

DETAILED DESCRIPTION:
People with a schizophrenia spectrum diagnosis often experience distressing worries or beliefs about other people intending to cause them harm (also known as paranoia). Paranoid beliefs are associated with significant distress and disruption to the person's life. This results in high use of services and costs to mental health providers.

The National Institute of Clinical Excellence recommends that cognitive behavioural therapy for psychosis (CBTp) is offered to everybody with a schizophrenia spectrum psychosis. The latest meta analyses report improved outcomes, and reduced inpatient stays following CBTp, making it a cost effective intervention.

Although improved outcomes have been obtained by therapies, CBTp has only small to moderate effects on paranoid beliefs. Further, training therapists to competently deliver CBTp is intensive, expensive and takes up to a year. CBTp is therefore not widely available to service users, resulting in inequalities in access to care.

The investigators are seeking to improve outcomes and accessibility of CBTp for people with distressing, paranoid beliefs. The proposed research programme aims to conduct a feasibility study of a brief therapeutic group intervention, aimed at targeting and improving anxiety processes which are causally implicated in paranoia.

The investigators have preliminary evidence indicating that the pilot intervention delivered in an individual format, with interactive multimedia content, reduced distressing beliefs and improved coping (Freeman et al, 2014). Participants also reported they found the interventions acceptable, enjoyable and useful. Based on these results, the investigators have further developed the intervention and the current study proposes to evaluate the modified intervention delivered in a group format. A pilot randomised controlled trial (RCT) of the novel group intervention will be conducted to inform its further development and to estimate key parameters required to plan a larger trial.

The feasibility and efficacy of the therapy will be investigated in a randomised controlled design (n = 35) with a between-groups longitudinal design to compare key outcomes between people who do and do not receive the intervention and to estimate key trial parameters. Participants will be randomised to either an immediate intervention or a delayed intervention condition (in which they are offered the intervention after completing all assessments) using a 2:1 ratio. Participants will be randomised after completing baseline measures using an independent web-based randomisation service. The researchers will be delivering the intervention and therefore will not be blind to group allocation. Participants will be recruited from community mental health teams and standalone psychology services in the South London and Maudsley NHS Foundation Trust.

As this is a pilot study, the statistical analysis will be mainly descriptive in nature, aiming to provide estimates of key trial parameters and to inform power calculations for a future larger scale trial. A description of the sample will be presented using means and standard deviations for continuous data, or medians and interquartile range if data are skewed. Frequencies and proportions will be used to analyse categorical variables. Feasibility of trial procedures will be assessed using proportions of predetermined parameters and their estimated 95% confidence intervals (CIs). Population variances for future power calculations will be determined using the upper 80th percentile of confidence intervals around the estimated population variance, as recommended by Browne (1995).

ELIGIBILITY:
Inclusion Criteria:

* Self reported worries about being harmed or at risk from others
* Non-affective psychosis(ICD10,F20-F29)
* Age 18-65
* Symptoms stable no major relapse or crisis in last 3 months prior to consent
* Sufficient command of English to provide informed consent, complete the measures and participate in the brief interventions
* Score above the cutoff for clinically significant levels of paranoia on the Green Paranoid Thoughts Scale (Green et al, 2008)
* Paranoia is triggered by being outside

Exclusion Criteria:

* Lack of capacity to provide informed consent
* Primary diagnosis of drug or alcohol use with secondary psychosis
* Primary diagnosis of mood disorder or bipolar affective disorder
* Primary diagnosis of learning difficulty
* Unstable residential arrangements (making a move away during the course of participation in the research likely)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Garety, CPsychol, MPhil, PhD, FBPsS, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, Psychology & Neuroscience (IoPPN), King's College London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Therapy | Delayed Therapy
Started | 13 | 5
Completed | 10 | 5
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Therapy | Delayed Therapy | Total
Number analyzed (Participants) | 13 | 5 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (10.4) | 46.6 (8.5) | 46.7 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 7 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 1 | 10
  Black | 2 | 4 | 6
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Green Paranoid Thoughts Scale (GPTS)
Description: The GPTS consists of two 16-item scales. Ideas of reference (part A) and ideas of persecution (part B) are rated over the past month on a scale ranging from one (not at all) to five (totally). A total score is produced by summing all items for part A and B (minimum score = 32; maximum score = 160). A higher score indicates more paranoid thoughts.
Time Frame: Assessed at baseline, at 6 weeks and 10 weeks
Population: A total of 18 participants were randomised. In the immediate therapy condition, 3 participants withdrew after baseline assessments and were not able to be contacted, 1 participant completed all assessments but did not feel able to attend the intervention. 1 participant was unable to complete all measures due to language difficulties and fatigue.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Therapy | Delayed Therapy
Number analyzed (Participants) | 10 | 5
score on a scale
  Baseline | 109.77 (13.18) | 114.6 (24.93)
  6 weeks (post therapy) | 84.8 (38.72) | 82.6 (30.25)
  10 weeks (follow up) | 82.1 (25.72) | 69 (36.22)

ADVERSE EVENTS:
Arm/Group | Immediate Therapy | Delayed Therapy
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/5
Other Adverse Events (participants affected / at risk) | 0/13 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No